CLINICAL TRIAL: NCT00451126
Title: Moderating Impact of Various Emotion Personality Factors on Salivary Cortisol
Brief Title: Moderating Impact of Various Emotion Personality Factors on Salivary Cortisol Response to a TSST
Acronym: cortpersonal
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Other Study IDs: personalityandcortisol
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Psychological Stress
Keywords: emotion; personality; social stress; appraisal
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With the aim of evaluating the putative impacts of emotion related personality factors on physical and mental disease and the mechanisms of these impacts, 58 students were submitted to a social stress test (Trier Social Stress Test) and salivary cortisol samples were taken. The subjects were also submitted to several personality trait inventory, that evaluated respectively Alexithymia, Emotional Intelligence, Resilience and the Five Factor Model of Personality.

The moderating impact of these factors on the cortisol response were analysed

ELIGIBILITY:
Inclusion Criteria:

* Students

Exclusion Criteria:

* Female,
* Smokers,
* Medication or alcohol abuse

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58
Dates: Start 2005-10; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luminet Olivier, PhD, Study Director — Fonds National de la Recherche Scientifique
Locations (1):
- Faculté de Psychologie, Université Catholique de Louvain, Louvain-la-Neuve, Belgium